CLINICAL TRIAL: NCT00459875
Title: Phase II Study of Sunitinib in Patients With Metastatic Papillary Renal Cell Carcinoma
Brief Title: Sunitinib in Treating Patients With Locally Recurrent or Metastatic Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-019; P30CA008748 (NIH); MSKCC-07019
Record Dates: First submitted 2007-04-11; First posted 2007-04-13 (Estimated); Results first posted 2015-11-26 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-10

CONDITIONS: Kidney Cancer
Keywords: recurrent renal cell cancer; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Sunitinib

ARMS (1):
- Sunitinib (Experimental): The treatment will include Sunitinib malate 50 mg self-administered orally, once daily in the evening, without regard to meals, for 4 consecutive weeks (28 days) followed by 2 weeks (14 days) off, to comprise a complete cycle of 6 weeks.
  Interventions: Drug: sunitinib malate

INTERVENTIONS:
Drug: sunitinib malate

SUMMARY:
RATIONALE: Sunitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well sunitinib works in treating patients with locally recurrent or metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of sunitinib malate in patients with locally recurrent or metastatic papillary renal cell carcinoma.

OUTLINE: Patients receive oral sunitinib malate once daily on days 1-28. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 28 days and every 2 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced renal cell carcinoma of papillary or other non-clear cell histology

  * Metastatic or locally recurrent disease
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral CT scan

  * The following are considered nonmeasurable disease:

    * Bone lesions
    * Ascites
    * Peritoneal carcinomatosis or miliary lesions
    * Pleural or pericardial effusions
    * Lymphangitis of the skin or lung
    * Cystic lesions
    * Irradiated lesions
* Patients with primary tumor in place who are eligible for surgery must have undergone prior partial or radical nephrectomy
* No history of or known brain metastases, spinal cord compression, or evidence of symptomatic brain or leptomeningeal carcinomatosis

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9.0 g/dL
* Calcium ≤ 12.0 mg/dL
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* AST and ALT ≤ 2.5 times ULN (5 times ULN if liver function abnormalities are due to underlying malignancy)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No hemorrhage ≥ grade 3 within the past 4 weeks
* No diagnosis of any second malignancy within the past 5 years, except for adequately treated basal cell carcinoma, squamous cell skin cancer, or in situ cervical cancer
* None of the following within the past 6 months:

  * Myocardial infarction
  * Severe or unstable angina
  * Coronary or peripheral artery bypass graft
  * Symptomatic congestive heart failure
  * Cerebrovascular accident or transient ischemic attack
  * Pulmonary embolism
* No ongoing cardiac dysrhythmias ≥ grade 2 or atrial fibrillation of any grade
* No prolongation of the QTc interval to > 450 msec (males) or > 470 msec (females)
* No uncontrolled hypertension (i.e., blood pressure > 150/100 mm Hg despite optimal medical therapy)
* No pre-existing thyroid abnormality, with thyroid function tests that cannot be maintained in the normal range with medication
* No known HIV or AIDS-related illness
* No other active infection
* No other severe acute or chronic medical or psychiatric condition or laboratory abnormality that would preclude study compliance

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior sunitinib malate
* Prior or concurrent bisphosphonates allowed
* More than 4 weeks since prior radiotherapy and recovered
* Prior palliative radiotherapy to metastatic lesions allowed provided there is ≥ 1 measurable lesion that has not been irradiated
* More than 4 weeks since prior major surgery and recovered
* No concurrent therapeutic doses of warfarin

  * Low-dose warfarin ≤ 2 mg daily for thromboprophylaxis allowed
  * Concurrent low molecular weight heparin for full anticoagulation allowed
* No other concurrent approved or investigational anticancer treatment, including chemotherapy, biological response modifiers, hormonal therapy, or immunotherapy
* No other concurrent investigational drugs
* No concurrent treatment on another clinical trial

  * Concurrent participation on supportive care trials or nontreatment trials (e.g., quality of life trials) allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-03; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Kroog, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Robert J. Motzer, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Molina AM, Feldman DR, Ginsberg MS, Kroog G, Tickoo SK, Jia X, Georges M, Patil S, Baum MS, Reuter VE, Motzer RJ. Phase II trial of sunitinib in patients with metastatic non-clear cell renal cell carcinoma. Invest New Drugs. 2012 Feb;30(1):335-40. doi: 10.1007/s10637-010-9491-6. Epub 2010 Aug 14. PMID 20711632

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib: The treatment will include Sunitinib malate 50 mg self-administered orally, once daily in the evening, without regard to meals, for 4 consecutive weeks (28 days) followed by 2 weeks (14 days) off, to comprise a complete cycle of 6 weeks.
  sunitinib malate
Period: Overall Study
Arm/Group | Sunitinib
Started | 24
Completed | 21
Not Completed | 3
Not completed — Ineligible participant | 1
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Sunitinib
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: Overall Objective Response Rate as Measured by RECIST
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 23
participants
  Partial Response (PR) | 1
  Stable Disease (SD) | 16
  Progression of Disease (POD) | 6

ADVERSE EVENTS:
Arm/Group | Sunitinib
Serious Adverse Events (participants affected / at risk) | 11/23
Other Adverse Events (participants affected / at risk) | 21/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib (N=23)
Coagulation, other (Blood and lymphatic system disorders) | 1 (1)
Creatinine (Blood and lymphatic system disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Fever (in the absence of neutropenia) (General disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Hemorrhage, Abdomen Not Otherwise Specified (NOS) (Gastrointestinal disorders) | 1 (1)
Nausea (General disorders) | 1 (1)
Pain - Abdomen NOS (General disorders) | 1 (1)
Pain - Back (General disorders) | 1 (1)
Pain - Other (specify) (General disorders) | 1 (1)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rigors/chills (General disorders) | 1 (1)
Thrombosis/thrombus/embolism (Cardiac disorders) | 2 (2)
Vomiting (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib (N=23)
ALT, SGPT (Blood and lymphatic system disorders) | 3 (3)
AST, SGOT (Blood and lymphatic system disorders) | 5 (5)
Bilirubin (hyperbilirubinemia) (Blood and lymphatic system disorders) | 3 (3)
Creatinine (Blood and lymphatic system disorders) | 3 (3)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 3 (3)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 4 (4)
Hemoglobin (Blood and lymphatic system disorders) | 9 (9)
Hypertension (Cardiac disorders) | 2 (2)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 10 (10)
Lymphopenia (Blood and lymphatic system disorders) | 5 (5)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 9 (9)
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 3 (3)
Platelets (Blood and lymphatic system disorders) | 6 (6)
Potassium, high (hyperkalemia) (Blood and lymphatic system disorders) | 6 (6)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 3 (4)
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 2 (2)
Thyroid function, high (Metabolism and nutrition disorders) | 5 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes